CLINICAL TRIAL: NCT03263000
Title: Study of the Photic Blink Reflex in Patients With Blepharospasm and Increased Blinking
Brief Title: Photic Blink Reflex in People With Blepharospasm and Increased Blinking
Status: Terminated | Type: Observational
Why Stopped: Protocol could not be carried out to achieve the aims of the study
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 170159; 17-N-0159
Record Dates: First submitted 2017-08-25; First posted 2017-08-28 (Actual); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Blepharospasm
Keywords: Belpharospasm; Blink Reflex; Eyeblink
MeSH Terms: conditions — Blepharospasm

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy: 24 healthy volunteers (HVs)
- Patients: 24 patients with blepharospasm
- Patients 2: 24 patients with increased blinking alone.

SUMMARY:
Background:

Some people who have increased blinking may later develop blepharospasm. Blepharospasm is a neurological disorder that causes involuntary closing of the eyes. Researchers want to learn more about how eyes close in response to different stimuli. They want to study this in healthy people, people with increased blinking, and people with blepharospasm.

Objective:

To learn how light exposure affects people with blepharospasm.

Eligibility:

People ages 18 and older with blepharospasm or increased blinking, and healthy volunteers

Design:

Participants will be screened with:

Medical history

Physical exam

Neurological exam

Participants will have up to 5 visits. The number of visits will depend on the number of tests they opt to have. They can opt to have up to 4 tests. Visits last 60-90 minutes. They cannot drink alcohol or caffeinated drinks for at least 12 hours before visits. Visits could include the following tests:

Evaluation of eyelid movements. This will be video recorded.

Electromyography: Small sticky electrodes are placed on the lower eyelid skin. These are attached to wires. Muscle activity is recorded during blink reflex procedures.

Electrical stimulation: An electrode is placed close to the eyebrow. It will deliver small electrical shocks. The strength of the shocks will be enough to provoke a blink.

Photic stimulation: A lamp is placed in front of the face. It will deliver single or paired flashes. The flashes will be at various intervals and intensities. Participants will wear a patch over one eye during this test.

Combination of electrical and photic stimulation

...

DETAILED DESCRIPTION:
Objective:

* The purpose of the first study of this protocol is to improve understanding of the role played by light sensitivity in the pathophysiology of blepharospasm (BPS).
* As a characteristic feature of BPS, the electrocutaneous blink reflex recovery cycle (EBR rc) shows an increased recovery index of R2 compared with healthy subjects.
* In the first study proposed under this protocol we will study the recovery cycle of the blink reflex evoked by a light stimulus (PBR rc) and the effect of a light stimulus on the EBR (MBR rc) in patient with BPS. Since photophobia and increased blinking are common symptoms in this group of patients, we will look for possible correlations between neurophysiological data and the Light Sensitivity Questionnaire (LSQ) or the Blink rate (Brt). The second study proposed under this protocol will explore the PBR rc and the MBR rc in patients with increased blinking alone, a condition indicated as a possible precursor of BPS.

Study population:

We plan to recruit 24 patients with blepharospasm, 24 healthy volunteers (HVs) and 24 patients with increased blinking alone.

Design:

In two different studies, we will compare all the results from the EBR rc, PBR rc and MBR rc between BPS patients (first study) or increased blinking patients (second study) and HVs. We will also look for possible correlation between the neurophysiologic data and the clinical scales acquired during a clinical assessment. In the EBR rc procedure, the supraorbital nerve will be stimulated with paired electrical stimuli at varying ISIs and the EMG response from the orbicularis oculi muscles will be recorded. In the PBR rc procedure, paired light stimuli will be given at varying interstimulus intervals (ISIs) and the EMG responses from the orbicularis oculi will be recorded. In the MBR rc study a weak light stimulation will be given at varying ISIs before an electrical stimulation of the supraorbital nerve. Each experimental procedure will last about 1 hour. There will be one screening visit and up to 4 testing visits per participant. However, participant can either undergo all the experimental procedures or participate in only some of them and will be allowed to participate in two experimental procedures per testing visit.

Outcome measurements:

* EBR rc, PBR rc, MBR rc: the electromyography (EMG) responses at different interstimulus intervals (ISIs).
* Blink rate: number of eye blinks per minute.
* LQs: the total score of the Light Questionnaire Scale.

These results will be compared between the two patient groups and HVs. We will look for possible correlations between neurophysiological and clinical data.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Must be 18 years or older
* For patients only: fulfill the criteria of

  * Primary BPS (either focal or related to segmental dystonia) in accordance with published criteria or
  * Excessive involuntary eyelid closure without sustained OO spasms in accordance with Conte et al + having a resting blink rate above 15 blinks per minute.
* Ability to give informed consent.
* Ability to comply with all study procedures.
* Agree to consume no caffeine or alcohol for 12 hours before participating in the testing visits.

EXCLUSION CRITERIA:

Any of the following will exclude PATIENTS from the study:

* Secondary causes of excessive involuntary eyelid closure such as ophthalmologist disorders involving the ocular surface, tear film, or eyelids.
* Any evidence suggesting a psychogenic movement disorder such as persisting unilateral or asymmetric symptoms, paroxysmal symptoms, and other inconsistencies such as pain, associated somatizations, blinking diminished by distraction, unusual sensory tricks, or unexpected response.
* Botulinum toxin treatment < 3 months prior to a testing visit.
* History of chronic exposure (>3 month) to dopamine receptor blocking agents before the onset of increased blinking alone or BPS.

Any of the following will exclude BOTH patients and healthy controls from the study:

* Has any major medical problem other than increased blinking or dystonia in patient groups (such as decompensated chronic diseases or conditions that cause serious disability such as congestive heart failure/NYHA score greater than or equal to 2, severe COPD, advanced neoplasia, severe arthritis, HIV/AIDS, blindness).
* Employees, staff or fellows of HMCS in NINDS.
* Has used illegal drugs within the past 6 months based on history. The intent is to exclude those with drug use that may affect study results.
* Self-reported consumption of more than 7 alcoholic drinks a week in the case of a woman and 14 alcoholic drinks a week in the case of a man.
* Abnormal findings on neurologic exam (other than increased blinking or dystonia in patient groups).
* Presence of anatomical or functional eyelid abnormalities other than involuntary eyelid closure or OOs spasms (including apraxia of eyelid opening, and other disorders such as tics or tardive syndromes).
* Has a neurologic disorder other than increased blinking or dystonia.
* Has major depression or any major mental disorders (axis I disorders).
* Has had a head injury where there was a loss of consciousness for more than a few seconds.
* Has a deep brain stimulator, pacemaker or other implantable electronic device subject to malfunction by electrical stimulation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We plan to recruit 24 patients with blepharospasm, 24 healthy volunteers (HVs) and 24 patients with increased blinking alone.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2017-10-30 (Actual); Primary Completion 2019-04-24 (Actual); Study Completion 2019-04-24 (Actual)

PRIMARY OUTCOMES:
Photic blink reflex recovery cycle | Single determination

SECONDARY OUTCOMES:
Electrocutaneous blink reflex recovery cycle; Blink rate; Light Questionnaire Scale | Single determination

CONTACTS AND LOCATIONS:
Overall Officials: Mark Hallett, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Adams WH, Digre KB, Patel BC, Anderson RL, Warner JE, Katz BJ. The evaluation of light sensitivity in benign essential blepharospasm. Am J Ophthalmol. 2006 Jul;142(1):82-87. doi: 10.1016/j.ajo.2006.02.020. PMID 16815254
- [Background] Albanese A, Bhatia K, Bressman SB, Delong MR, Fahn S, Fung VS, Hallett M, Jankovic J, Jinnah HA, Klein C, Lang AE, Mink JW, Teller JK. Phenomenology and classification of dystonia: a consensus update. Mov Disord. 2013 Jun 15;28(7):863-73. doi: 10.1002/mds.25475. Epub 2013 May 6. PMID 23649720
- [Background] Aramideh M, Eekhof JL, Bour LJ, Koelman JH, Speelman JD, Ongerboer de Visser BW. Electromyography and recovery of the blink reflex in involuntary eyelid closure: a comparative study. J Neurol Neurosurg Psychiatry. 1995 Jun;58(6):692-8. doi: 10.1136/jnnp.58.6.692. PMID 7608667